CLINICAL TRIAL: NCT05673629
Title: A Phase III, Open-label, Randomized, Controlled Study of Utidelone in Combination With AC Versus Docetaxel in Combination With AC for Neoadjuvant Chemotherapy in Patients With High-risk Early-stage or Locally Advanced HER2-negative Breast Cancer
Brief Title: Utidelone in Combination With AC Versus Docetaxel in Combination With AC for Neoadjuvant Chemotherapy in Patients With HER2-negative Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG01-2102
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The treatment group-Utidelone in combination with AC (Experimental): Utidelone Injection at 30 mg/m2/d administered on days 1-5 of each cycle. Doxorubicin Injection at 50mg/m2 and Cyclophosphamide Injection at 500 mg/m2 administered once daily on day 1 of each cycle.
  One treatment cycle has 21 days, and there are 6 cycles in total.
  Interventions: Drug: Utidelone Injection in combination with AC
- The control group-Docetaxel in combination with AC (Active Comparator): Docetaxel Injection at 75 mg/m2, Doxorubicin Injection at 50 mg/m2, and Cyclophosphamide Injection at 500mg/m2, administered on day 1 of each cycle.
  One cycle has 21 days, and there are 6 cycles in total.
  Interventions: Drug: Docetaxel Injection in combination with AC

INTERVENTIONS:
Drug: Utidelone Injection in combination with AC — The treatment group will be treated with Utidelone Injection at 30 mg/m2/d administered intravenously once daily on days 1-5 of each cycle, and Doxorubicin Injection at 50mg/m2 and Cyclophosphamide Injection at 500 mg/m2, administered intravenously respectively once daily on day 1 of each cycle. One treatment cycle has 21 days, and there are 6 cycles in total.
  After the neoadjuvant therapy, all patients suitable for surgery will have the operation, and they will be evaluated pre-operatively for clinical remission according to RECIST 1.1. For patients unsuitable for surgery, they will receive other treatments according to the clinical practice at each site.
  Safety evaluation will be performed 28 days after the last dose, and patients will be followed up for at least 3 years for disease recurrence.
  Arms: The treatment group-Utidelone in combination with AC
Drug: Docetaxel Injection in combination with AC — The control group will be treated with Docetaxel Injection at 75 mg/m2, Doxorubicin Injection at 50 mg/m2, and Cyclophosphamide Injection at 500mg/m2, administered intravenously once on day 1 of each cycle. One cycle has 21 days, and there are 6 cycles in total.
  After the neoadjuvant therapy, all patients suitable for surgery will have the operation, and they will be evaluated pre-operatively for clinical remission according to RECIST 1.1. For patients unsuitable for surgery, they will receive other treatments according to the clinical practice at each site.
  Safety evaluation will be performed 28 days after the last dose, and patients will be followed up for at least 3 years for disease recurrence.
  Arms: The control group-Docetaxel in combination with AC

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Utidelone plus AC versus Docetaxel plus AC as neoadjuvant chemotherapy in high-risk HER2-negative early-stage or locally advanced breast cancer.

In this phase III, multi-center, open-label, randomized controlled study, 552 subjects will be enrolled and randomly assigned in a 1:1 ratio to either the Utidelone plus AC group or the docetaxel plus AC group, stratified by hormone receptor status (ER and/or PgR positive vs ER and PgR negative).

DETAILED DESCRIPTION:
The subjects in treatment group will be treated with Utidelone at 30 mg/m2/d administered intravenously once daily on days 1-5 of each cycle, and doxorubicin at 50mg/m2 and cyclophosphamide at 500 mg/m2, administered intravenously once daily on day 1 of each cycle. One treatment cycle has 21 days, and there are in total 6 cycles. The subjects in control group will be treated with docetaxel at 75 mg/m2, doxorubicin at 50 mg/m2, and cyclophosphamide at 500mg/m2, administered intravenously once on day 1 of each cycle. One cycle has 21 days, and there are 6 cycles in total.

After the neoadjuvant therapy, all patients suitable for surgery should take the operation, and patients will be evaluated pre-operatively for clinical remission according to RECIST 1.1. After the surgery, patients will be evaluated for pathological remission, and physicians will recommend, according to clinical practice guidelines and clinical practice at each site, radiotherapy or adjuvant therapy for patients with corresponding clinical indications, and endocrine therapy for ER positive and/or PgR positive patients. Patients unsuitable for surgery receive other treatments according to the clinical practice at each site.

Safety evaluation will be performed 28 days after the last dose, and patients will be followed up for at least 3 years for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients who will receive initial treatment, 18 ≤ years of age ≤70.
2. Pathologically confirmed HER2-negative breast cancer at each investigational site with IHC at 0 or 1+, or IHC at 2+ with HER2 being negative by ISH (please refer to the ASCO/CAP Guideline 2020 for the relevant definition).
3. For patients with triple negative breast cancer, the requirement is tumor size>2 cm or lymph node-positive (T1, N1-3, M0, T2-4, any N, M0; tumor stage: II or III).
4. For patients with HR-positive and HER2-negative breast cancer, the requirement is (T2-4, N1-3, M0 or T2-4, N0 with high risk factors, M0):

   * Tumor size>2cm
   * lymph node-positive or high-risk factor with pathologically negative lymph node. High risk factors include:

   A. histologic grade 3.

   B. high Ki67 expression (≥20%).
5. Baseline routine blood tests within 1 week prior to enrollment is normal, with CTCAE grade ≤1 (based on normal values at each site's laboratory). No rhG-CSF use and no blood transfusion/EPO etc. within 14 days prior to enrollment.

   A. White blood cell count ≥ 4.0× 109/L;

   B. Neutrophil count ≥ 1.5 × 109/L;

   C. Platelet count ≥ 100 × 109/L;

   D. Hemoglobin ≥100 g/L.
6. Blood biochemistry test result is normal within 1 week prior to enrollment, with CTCAE grade ≤1 (based on normal values at each site's laboratory).

   A. Total bilirubin ≤ upper limit of normal (ULN).

   B. AST and ALT ≤ 1.5 x ULN.

   C. alkaline phosphatase ≤ 2.5×ULN.

   D. Serum creatinine ≤ 1.5×ULN.
7. Left ventricular ejection fraction (LVEF) on cardiac ultrasound ≥55%.
8. ECOG performance status 0 or 1.
9. Females of childbearing potential must agree to use effective contraception during the study and within 6 months after the last dose. The blood or urine pregnancy test for female patients of childbearing age prior to enrollment must be negative.
10. The patient willingly participates in this study, will sign the informed consent form, and commits to following the treatment and follow-up schedule.

Exclusion Criteria:

1. Stage IV metastatic breast cancer.
2. Inflammatory breast cancer.
3. Bilateral primary breast cancer (including invasive cancer and carcinoma in situ).
4. Patients who have previously received anti-tumor treatment or radiotherapy for any malignancy, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin and squamous cell carcinoma.
5. Patients who receive any sex hormone therapy (e.g., birth control pills, hormone replacement therapy, etc.), or any hormonal drug (e.g., raloxifene, tamoxifen, or other selective estrogen receptor modulators) for osteoporosis or breast cancer prevention.
6. Patients received major surgical operation unrelated to breast cancer within 4 weeks prior to randomization or having not yet fully recovered.
7. Patients with symptomatic peripheral neuropathy with CTCAE 5.0 grade ≥ 2.
8. Patients with severe cardiovascular diseases, including but not limited to:

   A. history of congestive heart failure or systolic dysfunction (LVEF < 50%).

   B. angina requiring anti-anginal medication.

   C. high-risk uncontrolled arrhythmias or severe conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second- to third-degree atrioventricular block, etc.; mean QTcF >470ms in 3 12-lead ECGs tests at rest.

   D. clinically significant heart valve disease with impaired cardiac function.

   E. Clinically uncontrollable hypertension.

   F. History of myocardial infarction.
9. Patients allergic to any ingredient of any drug to be administered in this study.
10. Patients unsuitable for corticosteroids.
11. Patients with active infection and currently in need of systemic anti-infective therapy.
12. Patients with history of immunodeficiency, including history of HIV, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation.
13. Patients who have participated in another interventional drug trial within 28 days prior to randomization or are concurrently participating in another clinical trial or using another investigational treatment.
14. Patients during pregnancy (positive pregnancy test), lactation.
15. Patients with any other co-morbidities that interfere with the regimens in this study, or in the opinion of the investigator, the subject has a history of other serious systemic disease or other reasons that make participation in this trial inadvisable.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients who will receive initial treatment, 18 ≤years of age ≤70.
Enrollment: 552 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Pathologic Complete Response | 24 months
  tpCR (ypT0/is, ypN0), percentage of patients with absence of invasive neoplastic cells in ipsilateral lymph nodes and the breast

SECONDARY OUTCOMES:
Breast Pathologic Complete Response | 24 months
  ypT0/is, percentage of patients whose pathological evaluation of hematoxylin and eosin-stained breast samples do not show any residual invasive carcinoma.
Objective Response Rate | 24 months
  Proportion of subjects who get to CR or PR during neoadjuvant therapy
3-year Event Free Survival | 36 months
  Event of interest, which included preoperative disease progression, postoperative disease recurrence, and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China